CLINICAL TRIAL: NCT07169071
Title: Effects of Expiratory Muscle Training in Children With Asthma: A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AtlasUmkaya05; 2023/10 (Other Grant/Funding Number: Istanbul Atlas University)
Record Dates: First submitted 2025-09-05; First posted 2025-09-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-09

CONDITIONS: Asthma Childhood; Respiratory Muscle Training
Keywords: Asthma; Expiratory Muscle Training
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Children in the experimental group will receive the same home-based chest physiotherapy program as the control group (8 weeks, 5 days per week, 30 minutes per day). In addition, they will perform expiratory muscle training (EMT) using a threshold device at 30% of their maximum expiratory pressure (MEP). EMT will be applied twice daily for 20 minutes, at least 5 days per week for 8 weeks. Resistance will be increased by 10% each week, adjusted according to tolerance and the presence of any complaints.
  Interventions: Other: Home-based chest physiotherapy program; Other: Expiratory Muscle Training
- Control group (Sham Comparator): Children in the control group will receive a home-based chest physiotherapy program for 8 weeks, 5 days per week, 30 minutes per day. The program will include breathing exercises, teaching of relaxation positions, cough training, breathing control strategies, and physical activity recommendations. In addition, participants will perform sham expiratory muscle training at the lowest fixed load, twice daily for 20 minutes, at least 5 days per week for 8 weeks.
  Interventions: Other: Home-based chest physiotherapy program

INTERVENTIONS:
Other: Home-based chest physiotherapy program — he program will include breathing exercises, teaching of relaxation positions, cough training, breathing control strategies, and physical activity recommendations.
Other: Expiratory Muscle Training — Participants perform expiratory muscle training (EMT) using a threshold device at 30% of their maximum expiratory pressure (MEP). The program consists of twice daily sessions, each lasting 20 minutes, at least 5 days per week, for 8 weeks. Resistance will be increased by 10% each week, adjusted according to tolerance and the presence of any complaints for experimental group.
  Arms: Experimental group

SUMMARY:
The goal of this randomized clinical trial is to evaluate the effectiveness of expiratory muscle training (EMT) as an adjunct to conventional chest physiotherapy in children with asthma. Respiratory muscle training has been shown to improve muscle strength, functional capacity, and symptom control in adults with asthma, but evidence in pediatric populations is limited, particularly regarding expiratory training. This study aims to determine whether adding EMT to standard physiotherapy enhances pulmonary function, respiratory muscle strength, asthma control, and functional capacity compared to chest physiotherapy alone. The main questions are: (1) Does EMT improve expiratory muscle strength and pulmonary function in children with asthma? (2) Does EMT contribute to better asthma control and overall physical performance? Participants will be randomly assigned to either conventional chest physiotherapy or chest physiotherapy plus EMT. Interventions will be delivered as a home-based, low-cost, feasible program, with training protocols standardized in terms of intensity, frequency, and duration.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8 and 18 years Clinically diagnosed with asthma Ability to walk, cooperate, and be clinically stable Willingness to participate in the study

Exclusion Criteria:

* History of hospitalization within the last 4 weeks prior to enrollment Hospitalization during the exercise training program Presence of secondary conditions that may affect respiratory function (e.g., kyphoscoliosis) Currently participating in or having participated in a regular exercise training program within the past year

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Respiratory Function Test | 8 weeks
  Change from baseline forced vital capacity (FVC) at 8 weeks.
Respiratory Function Test | 8 weeks
  Change from baseline forced forced expiratory volume in 1 (FEV1) second at 8 weeks.
Respiratory Function Test | 8 weeks
  Change from baseline peak expiratory flow (PEF) at 8 weeks.
Respiratory Function Test | 8 weeks
  Change from baseline FEV1/FVC at 8 weeks.
Respiratory Muscle Strength | 8 weeks
  Change from baseline maximum inspiratory pressure (MIP) at 8 weeks.
Respiratory Muscle Strength | 8 weeks
  Change from baseline maximum expiratory pressure (MEP) at 8 weeks.
Peripheral Muscle Strength | 8 weeks
  Change from baseline m. quadriceps strength at 8 weeks.
Functional Capacity | 8 weeks
  Change from baseline distance covered in six minute walk test at 8 weeks.
Peak Cough Flow | 8 weeks
  Change from baseline peak cough flow at 8 weeks.

SECONDARY OUTCOMES:
Asthma Control | 8 weeks
  Change from baseline Asthma Control Test at 8 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No